CLINICAL TRIAL: NCT04101188
Title: Mechanisms Underlying the Protective Vascular Effects of Dietary Potassium in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1472577
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Risk Factor
Keywords: Dietary Potassium; Dietary Sodium; Vascular Health

STUDY DESIGN:
Intervention Model Description: All participants will complete each arm. It is a crossover, randomized design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate Potassium/Low Sodium (Experimental): Subjects will be provided with a diet that is moderate in potassium and low in sodium.
  Interventions: Other: Moderate Potassium/Low Sodium Diet
- Moderate Potassium/High Sodium (Experimental): Subjects will be provided with a diet that is moderate in potassium and high in sodium.
  Interventions: Other: Moderate Potassium/High Sodium Diet
- High Potassium/High Sodium (Experimental): Subjects will be provided with a diet that is high in both potassium and sodium.
  Interventions: Other: High Potassium/High Sodium Diet

INTERVENTIONS:
Other: Moderate Potassium/Low Sodium Diet — Consumption of 10 days of a diet moderate in potassium and low in sodium.
  Arms: Moderate Potassium/Low Sodium
Other: Moderate Potassium/High Sodium Diet — Consumption of 10 days of a diet moderate in potassium and high in sodium.
  Arms: Moderate Potassium/High Sodium
Other: High Potassium/High Sodium Diet — Consumption of 10 days of a diet high in potassium and high in sodium.
  Arms: High Potassium/High Sodium

SUMMARY:
Americans continue to consume high amounts of sodium. Potassium is notable for its blood pressure lowering effects but less is known regarding its effect on the vasculature. This investigation seeks to determine the role of dietary potassium on the vasculature in the presence of a high sodium diet in salt-resistant adults.

DETAILED DESCRIPTION:
Significant public health efforts have been made towards salt reduction but most have met with failure. Dietary factors such high sodium/low potassium diets contribute to the development of cardiovascular diseases (CVDs) such as atherosclerosis and high blood pressure (BP). This is important as CVD is the number one killer in the U.S. While the role of these two nutrients on BP is widely accepted, their impact on the vasculature has received less attention. Endothelial dysfunction, characterized by impaired dilation, is an important non-traditional risk factor for atherosclerosis. Evidence supporting potassium's beneficial role on vascular health remains unclear although it may be more effective in the presence of a high sodium diet. A purported mechanism responsible for sodium-induced vascular dysfunction is overproduction of reactive oxygen species (ROS) resulting in reduced nitric oxide (NO) production/bioavailability. Additionally, high sodium diets have been shown to stiffen the endothelium. This investigation will evaluate the vascular effects of dietary potassium during a high salt diet including its impact on sodium-induced oxidative stress and endothelial cell stiffness.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* normal blood pressure
* normal resting ECG

Exclusion Criteria:

* hypertension
* history of heart disease
* diabetes
* kidney disease
* obese (BMI ≥30)
* significant weight changes in the last 6 months
* use of tobacco products
* pregnant
* on a special diet (gluten free; vegan)
* take any medications for the above conditions
* endurance trained athletes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Conduit artery endothelial-dependent dilation | on day 10 of the diet
  The change in flow-mediated dilation (FMD) between the 3 diets as assessed by brachial artery FMD
Microvascular function | on day 10 of the diet
  Cutaneous microvascular dilatory response to local heating assessed by laser Doppler flowmetry coupled with intradermal microdialysis

SECONDARY OUTCOMES:
Ambulatory BP monitoring | on day 7 and 10 of diet
  assessed by 24-hour ambulatory blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Shannon L Lennon, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided